CLINICAL TRIAL: NCT03517059
Title: Prospective Study of Dysarthria, and the Appearance of Non-dopaminergic Signs in Idiopathic PARKinson's Disease
Brief Title: Study of Dysarthria, and the Appearance of Non-dopaminergic Signs in Idiopathic PARKinson's Disease
Acronym: Prodygi-II
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_89; 2016-A01544-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
Keywords: Levodopa; axial symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD patients: 30 PD patients in ON and OFF levodopa conditions
- Healthy control subjects: 30 age matched healthy control subjects
- Neurological control subjects: 10 patients with defined supra nuclear palsy

SUMMARY:
Pilot study:

* Longitudinal follow up of the PRODY-GI cohort for parkinson's disease (PD)
* Observational study of upper and lower axial symptoms' occurence in 30 PD patients in on and off drug conditions, 30 aged matched control subjects and 10 control subjects with supra nuclear palsy
* Multi modal approach: functional MRI, clinical , ENT assessment, respiratory assessment, neuropsychological and gait evaluations

DETAILED DESCRIPTION:
Prospective, clinical assessment of :

* Cognition and diadochokinetic task during fMRI in 30 PD patients (in off and on condition)
* Motor assessment using VICON gait and balance analysis
* Pulmonary functional testing in OFF and ON drug condition
* Quality of life
* Clinical neurological MDS UPDRS , N Fog questionnaire
* ENT and speech therapist evaluation in OFF and ON drug condition

ELIGIBILITY:
Inclusion Criteria:

Parkinson's Disease group :

Patients with Parkinson's Disease, who where included in the PRODYGI-1 cohort still meeting the MP criteria, Always followed in the service of neurology and pathology of the movement.

Pathological control group:

* Patients suffering from Richardson syndrome.
* Aged over 18

Healthy control group:

* Age-matched (± 5 years)
* Recruited on the basis of volunteering.
* free from any progressive neurological pathology after clinical examination and MoCA.

Exclusion Criteria:

For all groups:

* Pregnant or lactating woman
* Extra-neurological severe respiratory pathology
* Terminal heart failure
* Contraindication to MRI
* Refusal / withdrawal / inability to give consent
* ENT pathology.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease (PD)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Change in the neural network between patients in OFF levodopa conditions and control subjects | Between two evaluation visits, on average at 3 months (baseline- 3 months)
  Measure evaluated by functional MRI during the realisation of a cognitive task: symbol digit modality test

SECONDARY OUTCOMES:
Change in the neural network between patients in OFF-drug conditions and healthy control subjects | Between two evaluation visits, on average at 3 months (baseline- 3 months)
  Measure evaluated by functional MRI during the realisation of two motor tasks
Change in the neural network between patients in OFF-drug conditions and healthy control subjects | Between two evaluation visits, on average at 3 months (baseline- 3 months)
  Measure evaluated by resting state functional MRI
Change in the neural network between OFF-drug condition and ON-drug condition in patients | Between two evaluation visits, on average at 3 months (baseline- 3 months)
  Measure evaluated by functional MRI, during the realisation of one cognitive task and two motor tasks
Change in the neural network between patients in OFF-drug conditions and neurological control subjects (with supra nuclear palsy) | Between two evaluation visits, on average at 3 months (baseline- 3 months)
  Measure evaluated by functional MRI, during the realisation of one cognitive task and two motor tasks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MOREAU, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No